CLINICAL TRIAL: NCT04150003
Title: Multicenter, Randomize Study to Evaluate the Effect of a Physical Training Structured Program After a Pulmonary Thromboembolism in the Restoration Lung Perfusion
Brief Title: Study on the Effect of a Physical Training Structured Program After a Pulmonary Thromboembolism
Acronym: TEP-RR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TEP-RR
Record Dates: First submitted 2019-10-22; First posted 2019-11-04 (Actual); Last update posted 2021-01-14 (Actual); Status verified 2021-01

CONDITIONS: Pulmonary Embolism
Keywords: Venous Thromboembolic Disease; Pulmonary Embolism; Rehabilitation program; Exercise training
MeSH Terms: conditions — Pulmonary Embolism | interventions — Rehabilitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pulmonary Rehabilitation program (Experimental): 10-weeks structured exercise-based intervention protocol on the restoration of lung blood flow after an acute PE
  Interventions: Behavioral: Pulmonary Rehabilitation program
- Usual care (Active Comparator): Protocolized usual care for patient suffering PE
  Interventions: Other: Usual care

INTERVENTIONS:
Behavioral: Pulmonary Rehabilitation program — Structured rehabilitation program of directed exercises
  Other Names: Rehabilitation program
  Arms: Pulmonary Rehabilitation program
Other: Usual care — Usual care for patients who had suffered a Pulmonary Embolism
  Arms: Usual care

SUMMARY:
Exercise training, as the core component of a Pulmonary Rehabilitation program, may help restore arterial blood flow in the lungs of patients who had suffered Pulmonary Embolism (PE), stimulating and promoting vasodilator effects, repairing the damaged endothelium and recruiting new blood vessels and also inducing a net fibrinolytic balance. Besides, exercise training could have a positive effect on quality of life of these patients.

DETAILED DESCRIPTION:
An experimental multicenter study is proposed , randomized according to parallel assignation and blinded to third ones to evaluate the effect of a 10-weeks structured exercise-based intervention protocol on the restoration of lung blood flow after an acute PE.

Main objective is to compare the efficacy and safety in terms of quantitative measures from lung scintigraphy, of lung perfusion versus usual care in patients with PE. Additionally the study is aimed to identify bio-markers of response to treatment (mRNAs, MPs and proteomic approach) and to analyze the effects of training on exercise capacity, quality of life parameters and anxiety depression scores.

ELIGIBILITY:
Inclusion Criteria:

Patients 18 years or older at PE diagnosis PE diagnosis confirmed by imaging tests according guidelines Patients under correct anticoagulant treatment Persistent Lung Perfusion Defects at one month after PE diagnosis. Signed Consent Inform

Exclusion Criteria:

Incidental or silent PE Pregnant or puerperal woman Life expectancy less than 6 months Severe comorbidities (NYHA 4 in severe heart failure; COPD, gold D; severe psychiatric illness) Any disability for physical exercise according to their doctors

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2021-11-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in the rate of lung perfusion defects after PE | Baseline up to one month after the episode of PE, final after 12 weeks of randomization
  Lung scintigraphy of lung perfusion

SECONDARY OUTCOMES:
Identification of biomarkers of response to treatment | The day the randomization occurs and the final visit after 12 weeks of the randomization
  Changes from baseline in the determination of mRNAs
Identification of another biomarkers of response to treatment | The day the randomization occurs and the final visit after 12 weeks of the randomization
  Changes from baseline in the determination of MPs (Microparticle (MP) Microparticles (MPs)
Change in the percent predicted peak oxygen uptake (VO2 peak) after PE | Baseline up to one month after the episode of PE, final after 12 weeks of randomization
  Peak Oxygen uptake (VO2 peak) is obtained from Cardiopulmonary Exercise Test
Change in the EuroQol scale | Baseline up to one month after the episode of PE, final after 12 weeks of randomization
  Visual analog score (0-100, lower score indicate worse outcome)
Change in the PEmb-QoL questionnaire by a PEmb-QoL - | "Baseline up to one month after the episode of PE, final after 12 weeks of randomization
  PEmb-QoL summary score (0-100, higher score indicate worse outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Remedios Otero, MD-PhD, Study Chair — Hospitales Universitarios Virgen del Rocío
Locations (3):
- Spain (3):
  - Hospital de Txagorritxu, Vitoria-Gasteiz, Alava
  - Hospital Universitario Virgen del Rocio, Seville, Andalusia
  - Hospital Universitario Virgen Macarena, Seville

IPD SHARING:
Plan to Share IPD: Yes
Results to be published in impact factor journals
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After the end of analysis and publication of results
Access Criteria: collaborators in the design and performance of the study